CLINICAL TRIAL: NCT02162719
Title: A Randomized, Phase II, Multi-Center, Placebo-Controlled Study of Ipatasertib (GDC-0068), an Inhibitor of Akt, in Combination With Paclitaxel as Front-Line Treatment for Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: A Study Assessing the Safety and Efficacy of Adding Ipatasertib to Paclitaxel Treatment in Participants With Breast Cancer That Has Spread Beyond the Initial Site, and the Cancer Does Not Have Certain Hormonal Receptors
Acronym: LOTUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO29227; 2014-000469-35 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ipatasertib + Paclitaxel (Experimental): Participants randomised to receive paclitaxel 80 mg/m^2, intravenously on Days 1, 8, and 15 along with ipatasertib 400 mg, orally, once daily from Days 1-21 in each cycle of 28 days until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Placebo + Paclitaxel (Placebo Comparator): Participants randomised to receive paclitaxel 80 mg/m^2, intravenously on Days 1, 8, and 15 along with placebo matching ipatasertib, orally, once daily from Days 1-21 in each cycle of 28 days until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Ipatasertib — Participants received ipatasertib orally 400 milligrams (mg) daily on Days 1-21 of each 28-day cycle.
  Other Names: GDC-0068
  Arms: Ipatasertib + Paclitaxel
Drug: Paclitaxel — Participants received paclitaxel 80 milligrams per square meter (mg/m^2) intravenously (IV) on Days 1, 8, and 15 of each cycle.
Drug: Placebo — Participants received oral placebo matched to ipatasertib, daily on Days 1-21 of each 28-day cycle.
  Arms: Placebo + Paclitaxel

SUMMARY:
This multicenter, randomized, double-blind study will estimate the efficacy, safety and tolerability of ipatasertib combined with paclitaxel compared with placebo combined with paclitaxel in participants with inoperable locally advanced or metastatic triple-negative breast cancer (mTNBC), as measured by progression-free survival (PFS) in all participants and in participants with phosphatase and tensin homolog (PTEN)-low tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented triple-negative adenocarcinoma of the breast that is inoperable locally advanced or metastatic and is not amenable to resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumor specimen, required prior to randomization
* Measurable disease, according to the RECIST v1.1
* Adequate hematologic and organ function within 14 days before the first study treatment
* For female participants of childbearing potential, agreement (by both participant and partner) to use an effective form of contraception for the duration of the study and for 6 months after last dose of study treatment

Exclusion Criteria:

* Any previous therapy, including chemotherapy or hormonal or targeted therapy, for inoperable locally advanced or metastatic triple-negative adenocarcinoma of the breast. Participants may have received prior neoadjuvant or adjuvant chemotherapy and/or radiation treatment for locally advanced triple negative adenocarcinoma, provided all treatments were completed greater than or equal to (>/=) 6 months prior to Cycle 1 Day 1. Locally recurrent disease must not be amenable to resection with curative intent
* Any radiation treatment to metastatic site within 28 days of Cycle 1, Day 1
* Known Human Epidermal Growth Factor Receptor 2 (HER2) positive, erythrocyte receptor (ER) positive, or progesterone receptor (PR) positive breast cancer
* Previous therapy with Akt, PI3K, and/or mTOR inhibitors
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Known presence of the brain or spinal cord metastasis, as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening or prior radiographic assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (17):
  - St Jude Heritage Medical Group, Fullerton, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cancer Care Assoc Med Group, Los Angeles, California
  - UCLA Medical Center, Santa Monica, California
  - Holycross Medical Group, Fort Lauderdale, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Carolinas Healthcare System, Charlotte, North Carolina
  - The WEST CLINIC, P.C., Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Northern Utah Associates, Ogden, Utah
  - Northwest Medical Specialties, Lakewood, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
- Sint Augustinus Wilrijk, Wilrijk, Belgium
- France (5):
  - Institut Bergonié Centre Régional de Lutte Contre Le Cancer de Bordeaux Et Sud Ouest, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - Clinique Armoricaine de Radiol, Saint-Brieuc
- Italy (3):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Istituto Nazionale dei Tumori; Divisione Oncologia Chirurgica e Ginecologica, Milan, Lombardy
  - Istituto Oncologico Veneto IRCCS Farmacia Ospedaliera, Padua, Veneto
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre, Singapore
- South Korea (6):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - MD Anderson Cancer Center, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Farmacia, Madrid
  - Hospital Virgen del Rocio, Seville
- Taiwan (4):
  - China Medical University Hospital, North Dist.
  - Chi Mei Medical Center, Yong kang; Endocrinology, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou; Dept of Surgery, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kim SB, Dent R, Im SA, Espie M, Blau S, Tan AR, Isakoff SJ, Oliveira M, Saura C, Wongchenko MJ, Kapp AV, Chan WY, Singel SM, Maslyar DJ, Baselga J; LOTUS investigators. Ipatasertib plus paclitaxel versus placebo plus paclitaxel as first-line therapy for metastatic triple-negative breast cancer (LOTUS): a multicentre, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2017 Oct;18(10):1360-1372. doi: 10.1016/S1470-2045(17)30450-3. Epub 2017 Aug 8. PMID 28800861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 44 centers in 8 countries.
Pre-assignment Details: A total of 166 participants were screened, out of which 42 participants failed screening. A total of 124 participants were enrolled at 44 sites. Results are reported here up to clinical cut-off date of 31st August 2019.
Groups:
- Ipatasertib and Paclitaxel: Participants randomised to receive paclitaxel 80 mg/m^2, intravenously on Days 1, 8, and 15 along with ipatasertib 400 mg, orally, once daily from Days 1-21 in each cycle of 28 days until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
- Placebo and Paclitaxel: Participants randomised to receive paclitaxel 80 mg/m^2, intravenously on Days 1, 8, and 15 along with placebo matching ipatasertib, orally, once daily from Days 1-21 in each cycle of 28 days until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
Period: Overall Study
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Started | 62 | 62
Completed | 0 | 0
Not Completed | 62 | 62
Not completed — Death | 41 | 46
Not completed — Lost to Follow-up | 1 | 3
Not completed — Disease Progression | 2 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Discontinuation of Overall Survival Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.4) | 54.4 (10.9) | 54.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 51 | 52 | 103
  Not Stated | 5 | 5 | 10
  Unknown | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 28 | 30 | 58
  Black or African American | 5 | 3 | 8
  White | 26 | 28 | 54
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined by investigator review of tumor assessments by RECIST, v1.1 or death on study (<=30 days after the last dose of study treatment regimen) from any cause, whichever occurred first.
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 07 June 2016)
Population: The Intent to treat (ITT) population was defined as all randomized participants allocated to the treatment arm to which they were randomized.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 62 | 62
Months | 6.18 (4.57) [4.57 to 7.33] | 4.93 (3.58) [3.58 to 5.36]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.0372, Log Rank — Stratification variables were adjuvant/neoadjuvant treatment including treatment with or without radiation, disease-free interval from last dose (<=12 vs >12 months vs. no prior chemotherapy), PTEN status of tumor (H-score 0, vs. 1 to 150, vs. >150); Hazard Ratio (Stratified Analysis) = 0.60, 90% CI 2-sided [0.40 to 0.91]

2. Primary Outcome: PFS in Participants With Phosphatase and Tensin Homolog (PTEN)-Low Tumors
Description: as for outcome 1
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 07 June 2016)
Population: The ITT population included all randomized participants allocated to the treatment arm to which they were randomized. Participants with PTEN-low tumors were evaluated for this endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 25 | 23
Months | 6.18 (3.65) [3.65 to 9.10] | 3.65 (2.53) [2.53 to 5.75]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.1753, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (Stratified Analysis) = 0.59, 90% CI 2-sided [0.30 to 1.16]

3. Secondary Outcome: PFS in Participants With Phosphatidylinositol-4,5-bisphosphate 3-kinase Catalytic Subunit Alpha (PIK3CA)/ Protein Kinase B (AKT1)/ PTEN-altered Tumors
Description: as for outcome 1
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 07 June 2016)
Population: The ITT population was defined as all randomized participants allocated to the treatment arm to which they were randomized. Participants with PIK3CA/AKT1/PTEN-altered tumors were evaluated for this endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 26 | 16
Months | 9.03 (4.57) [4.57 to 12.88] | 4.93 (3.58) [3.58 to 5.39]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.3636, Log Rank; Hazard Ratio (Unstratified Analysis) = 0.76, 90% CI 2-sided [0.46 to 1.27]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 31 August 2019)
Population: The ITT population was defined as all randomized participants allocated to the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 62 | 62
months | 25.8 (18.6) [18.6 to 28.6] | 16.9 (14.6) [14.6 to 24.6]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.3607, Log Rank — Stratification variables were adjuvant/neoadjuvant treatment including treatment with/without radiation, disease-free interval from last dose (<=12 vs >12 months vs. no prior chemotherapy), PTEN status of tumor (H-score 0, vs. 1 to 150, vs. >150); Hazard Ratio (Stratified Analysis) = 0.80, 95% CI 2-sided [0.50 to 1.28]

5. Secondary Outcome: OS in Participants With PTEN-Low Tumors
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 31 August 2019)
Population: The ITT population was defined as all randomized participants allocated to the treatment arm to which they were randomized. Participants with PTEN-low tumors were evaluated for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 25 | 23
months | 23.1 (18.3) [18.3 to 28.6] | 15.8 (9.0) [9.0 to 29.1]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.4422, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (Stratified Analysis) = 0.73, 95% CI 2-sided [0.32 to 1.65]

6. Secondary Outcome: OS in Participants With PIK3CA/AKT1/PTEN-altered Tumors
Description: OS was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline up to 30 days after the last dose of study drug administration (Clinical Cut Off Date: 31 August 2019)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 26 | 16
months | 25.8 (18.6) [18.6 to 35.2] | 22.1 (8.7) [8.7 to 999]
Statistical Analysis 1: Comparison: Ipatasertib and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority; p = 0.7599, Log Rank; Hazard Ratio (Unstratified Analysis) = 1.13, 95% CI 2-sided [0.52 to 2.47]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: Confirmed tumor ORR in participants with measurable disease at baseline was assessed by the investigator per RECIST, v1.1. Confirmed ORR was defined as the percentage of participants who achieved either a complete response or partial response based on the investigator assessment that was confirmed by a repeat assessment no less than 4 weeks after the criteria for response was first met. Participants for whom no records of post-baseline tumor assessments were reported were counted as non-responders. Complete response (CR): disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 62 | 62
Percentage of Participants | 40.3 (30.64) [30.64 to 50.90] | 32.3 (23.35) [23.35 to 42.36]

8. Secondary Outcome: ORR in Participants With PTEN-Low Tumors
Description: as for outcome 7
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 25 | 23
Percentage of Participants | 48.0 (30.73) [30.73 to 64.00] | 26.1 (12.02) [12.02 to 43.12]

9. Secondary Outcome: ORR in Participants With PIK3CA/AKT1/PTEN-altered Tumors
Description: Confirmed tumor ORR in subjects with measurable disease at baseline was assessed by the investigator per RECIST, v1.1. Confirmed ORR was defined as the percentage of subjects who achieved either a complete response or partial response based on the investigator assessment that was confirmed by a repeat assessment no less than 4 weeks after the criteria for response was first met. Subjects for whom no records of post-baseline tumor assessments were reported were counted as non-responders. Complete response (CR): disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 26 | 16
Percentage of Participants | 50.0 (34.24) [34.24 to 65.76] | 43.8 (23.53) [23.53 to 66.66]

10. Secondary Outcome: Duration of Response
Description: Duration of objective response in subjects with measurable disease at baseline was defined as the time from first observation of an objective tumor response until first observation of disease progression, as assessed by the investigator per modified RECIST, v1.1.
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: The ITT population was defined as all randomized participants allocated to the treatment arm to which they were randomized. Only participants who achieved a confirmed objective response were included in the analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 25 | 20
months | 7.85 [5.65 to NA] — Upper Limit of Duration of Response was not reached due to low number of participants with events. | 7.43 [3.88 to 9.20]

11. Secondary Outcome: Duration of Response in Participants With PTEN-Low Tumors
Description: as for outcome 10
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: ITT population included all randomized participants allocated to the treatment arm to which they were randomized. Participants with PTEN-low tumors were evaluated for this endpoint. Only participants who achieved a confirmed objective response were included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 12 | 6
Months | 6.54 [4.44 to NA] — Upper Limit of Duration of Response was not reached due to low number of participants with events. | 7.49 [7.29 to NA] — Upper Limit of Duration of Response was not reached due to low number of participants with events.

12. Secondary Outcome: Duration of Response in Participants With PIK3CA/AKT1/PTEN-altered Tumors
Description: Duration of objective response in participants with measurable disease at baseline was defined as the time from first observation of an objective tumor response until first observation of disease progression, as assessed by the investigator per modified RECIST, v1.1.
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: ITT population included all randomized participants allocated to the treatment arm to which they were randomized. Participants with PIK3CA/AKT1/PTEN-altered tumors were evaluated for this endpoint. Only participants who achieved a confirmed objective response were included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 13 | 7
Months | 11.24 [5.59 to NA] — Upper Limit of Duration of Response was not reached due to low number of participants with events. | 6.06 [3.78 to 7.56]

13. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from randomization to the first occurrence of disease progression, as determined by investigator review of tumor assessments by RECIST, v1.1.
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: ITT population included all randomized participants allocated to the treatment arm to which they were randomized.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 62 | 62
Months | 6.18 (4.57) [4.57 to 7.33] | 4.96 (3.61) [3.61 to 5.39]

14. Secondary Outcome: Time to Disease Progression in Participants With PTEN-Low Tumors
Description: as for outcome 13
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: ITT population included all randomized participants allocated to the treatment arm to which they were randomized. Participants with PTEN low tumors were evaluated for this endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 25 | 23
Months | 6.18 (3.65) [3.65 to 9.10] | 3.94 (2.53) [2.53 to 7.33]

15. Secondary Outcome: Time to Disease Progression in Participants With PIK3CA/AKT1/PTEN-altered Tumors
Description: as for outcome 13
Time Frame: Baseline up to every 8 weeks until documented disease progression (Clinical Cut Off Date: 07 June 2016)
Population: ITT population included all randomized participants allocated to the treatment arm to which they were randomized. Participants with PIK3CA/AKT1/PTEN-altered tumors were evaluated for this endpoint.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 26 | 16
Months | 9.03 (4.57) [4.57 to 12.88] | 4.93 (3.58) [3.58 to 5.39]

16. Secondary Outcome: Safety: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to 30 days after the last dose of study drug or until initiation of another anti-cancer therapy, whichever occurs first (up to 3 years, 3 months)
Population: The Safety population included all treated participants with participants allocated to the treatment arm associated with the regimen that they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 61 | 62
Percentage of Participants | 100.0 | 96.8

17. Secondary Outcome: Pharmacokinetic Endpoint: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to 24 Hours (AUC0-24h) of Ipatasertib
Description: PK parameters were not calculated due to sparse PK sampling.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 8
Population: The PK Analysis population was defined as all participants who had evaluable PK data.
Measure: Number; unit: h*ng/mL/mg
Arm/Group | Ipatasertib and Paclitaxel
Number analyzed (Participants) | 61
h*ng/mL/mg | NA — Due to sparse PK sampling.

18. Secondary Outcome: Pharmacokinetic Endpoint: Apparent Clearance Following Oral Dosing (CL/F) of Ipatasertib
Description: PK parameters were not calculated due to sparse PK sampling.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 8
Population: The PK Analysis population was defined as all participants who had evaluable PK data.
Measure: Number; unit: ml/hr
Arm/Group | Ipatasertib and Paclitaxel
Number analyzed (Participants) | 61
ml/hr | NA — Due to sparse PK sampling.

19. Secondary Outcome: Patient Reported Outcome (PRO) Measure: Mean Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30-item (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30 included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), single items (dyspnoea, appetite loss, insomnia, constipation/diarrhea, financial difficulties). Most questions used 4-point scale (1=Not at all to 4=Very much; 2 questions used 7-point scale [1=very poor to 7=Excellent]). Scores averaged, transformed to 0-100 scale; a higher score=better level of functioning. For symptom scale scores, higher level=severe level of symptoms. "A change of at least 10 points from baseline is considered clinically meaningful (Osoba D, Rodrigues G, Myles J, et al. Interpreting the significance of changes in health-related quality of life score. J Clin Oncol 1998;16:139-44). PRO measures were analyzed from baseline up to cycle 5. Scores from later timepoints were not analyzed due to attrition (in both arms, fewer than 50% of participants remained on treatment beyond cycle 5).
Time Frame: Baseline (Cycle 1 Day 1) up to Cycle 5 Day 1
Population: The PRO Analysis population was defined as the ITT population with a baseline and at least one post baseline PRO assessment. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 57 | 53
unit on a scale
  Appetite loss:Cycle 2 | 7.60 (28.18) | -0.63 (24.88)
  Appetite loss:Cycle 3: number analyzed (Participants) | 46 | 43
  Appetite loss:Cycle 3 | 9.42 (21.84) | -3.88 (24.35)
  Appetite loss:Cycle 4: number analyzed (Participants) | 49 | 40
  Appetite loss:Cycle 4 | 5.44 (23.91) | -4.17 (25.25)
  Appetite loss:Cycle 5: number analyzed (Participants) | 35 | 30
  Appetite loss:Cycle 5 | 0.00 (18.08) | -1.11 (25.50)
  Cognitive Functioning: Cycle 2 Day 1 | 1.17 (14.04) | 0.63 (17.28)
  Cognitive Functioning: Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Cognitive Functioning: Cycle 3 Day 1 | -1.81 (19.64) | -1.81 (19.64)
  Cognitive Functioning: Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Cognitive Functioning: Cycle 4 Day 1 | -3.40 (15.95) | 0.00 (20.32)
  Cognitive Functioning: Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Cognitive Functioning: Cycle 5 Day 1 | 0.00 (13.80) | -4.44 (19.54)
  Constipation: Cycle 2 Day 1 | 5.85 (24.50) | 0.63 (25.73)
  Constipation: Cycle 3 Day 1: number analyzed (Participants) | 46 | 42
  Constipation: Cycle 3 Day 1 | 2.90 (19.66) | 1.59 (22.03)
  Constipation: Cycle 4 Day 1: number analyzed (Participants) | 48 | 40
  Constipation: Cycle 4 Day 1 | 1.39 (16.78) | 0.83 (30.65)
  Constipation: Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Constipation: Cycle 5 Day 1 | 2.78 (14.64) | 1.11 (20.50)
  Diarrhoea: Cycle 2 Day 1 | 17.54 (30.28) | 1.89 (15.21)
  Diarrhoea: Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Diarrhoea: Cycle 3 Day 1 | 23.91 (34.90) | 3.88 (18.13)
  Diarrhoea: Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Diarrhoea: Cycle 4 Day 1 | 19.73 (34.64) | 0.83 (15.99)
  Diarrhoea: Cycle 5 Day 1: number analyzed (Participants) | 35 | 30
  Diarrhoea: Cycle 5 Day 1 | 21.90 (37.87) | 1.11 (16.34)
  Dyspnea: Cycle 2 Day 1: number analyzed (Participants) | 57 | 52
  Dyspnea: Cycle 2 Day 1 | 2.92 (19.19) | 0.00 (18.67)
  Dyspnea: Cycle 3 Day 1: number analyzed (Participants) | 46 | 41
  Dyspnea: Cycle 3 Day 1 | 5.07 (23.27) | 2.44 (22.84)
  Dyspnea: Cycle 4 Day 1: number analyzed (Participants) | 49 | 39
  Dyspnea: Cycle 4 Day 1 | 3.40 (25.68) | 5.13 (22.35)
  Dyspnea: Cycle 5 Day 1: number analyzed (Participants) | 36 | 28
  Dyspnea: Cycle 5 Day 1 | 5.56 (25.82) | 4.76 (23.51)
  Emotional Functioning: Cycle 2 Day 1 | 12.09 (15.90) | 4.72 (16.87)
  Emotional Functioning: Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Emotional Functioning: Cycle 3 Day 1 | 7.37 (17.18) | 3.88 (20.36)
  Emotional Functioning: Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Emotional Functioning: Cycle 4 Day 1 | 8.22 (16.53) | 2.71 (21.47)
  Emotional Functioning: Cycle 5 Day 1: number analyzed (Participants) | 35 | 30
  Emotional Functioning: Cycle 5 Day 1 | 8.73 (16.30) | 1.39 (17.79)
  Fatigue: Cycle 2 Day 1 | 7.99 (22.69) | -1.36 (16.98)
  Fatigue: Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Fatigue: Cycle 3 Day 1 | 9.18 (22.63) | 1.42 (19.44)
  Fatigue: Cycle 4 Day 1: number analyzed (Participants) | 49 | 39
  Fatigue: Cycle 4 Day 1 | 7.94 (20.91) | 1.85 (21.64)
  Fatigue: Cycle 5 Day 1: number analyzed (Participants) | 35 | 30
  Fatigue: Cycle 5 Day 1 | 10.32 (20.35) | 1.67 (20.59)
  Financial difficulties Cycle 2 Day 1: number analyzed (Participants) | 56 | 52
  Financial difficulties Cycle 2 Day 1 | 3.57 (21.72) | 0.00 (20.87)
  Financial difficulties Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Financial difficulties Cycle 3 Day 1 | 0.72 (22.76) | -3.88 (24.35)
  Financial difficulties Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Financial difficulties Cycle 4 Day 1 | 3.40 (23.81) | -0.83 (29.71)
  Financial difficulties Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Financial difficulties Cycle 5 Day 1 | 2.78 (25.67) | 1.11 (26.96)
  Nausea/Vomiting Cycle 2 Day 1 | 9.06 (19.43) | 2.83 (15.24)
  Nausea/Vomiting Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Nausea/Vomiting Cycle 3 Day 1 | 6.52 (14.26) | 3.10 (14.21)
  Nausea/Vomiting Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Nausea/Vomiting Cycle 4 Day 1 | 6.80 (17.32) | 3.75 (17.50)
  Nausea/Vomiting Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Nausea/Vomiting Cycle 5 Day 1 | 3.70 (7.03) | 0.00 (23.16)
  Pain Cycle 2 Day 1 | -3.80 (22.93) | -7.86 (23.02)
  Pain Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Pain Cycle 3 Day 1 | -4.71 (26.45) | -7.36 (26.80)
  Pain Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Pain Cycle 4 Day 1 | 1.36 (28.63) | -3.33 (31.62)
  Pain Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Pain Cycle 5 Day 1 | 0.00 (26.13) | -5.56 (25.27)
  Physical Functioning Cycle 2 Day 1 | -4.53 (14.23) | -0.16 (12.96)
  Physical Functioning Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Physical Functioning Cycle 3 Day 1 | -5.94 (15.54) | -1.71 (13.88)
  Physical Functioning Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Physical Functioning Cycle 4 Day 1 | -9.12 (13.92) | -3.17 (16.54)
  Physical Functioning Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Physical Functioning Cycle 5 Day 1 | -8.56 (13.47) | -4.44 (14.26)
  Global health status Cycle 2 Day 1 | -4.68 (22.33) | 4.72 (18.38)
  Global health status Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Global health status Cycle 3 Day 1 | -8.15 (21.55) | 3.29 (21.37)
  Global health status Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Global health status Cycle 4 Day 1 | -8.50 (21.62) | -1.46 (26.61)
  Global health status Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Global health status Cycle 5 Day 1 | -6.48 (22.55) | -5.00 (21.62)
  Role Functioning Cycle 2 Day 1 | -5.85 (20.04) | 0.63 (22.40)
  Role Functioning Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Role Functioning Cycle 3 Day 1 | -10.51 (24.43) | -2.71 (22.69)
  Role Functioning Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Role Functioning Cycle 4 Day 1 | -13.95 (25.76) | -6.25 (26.34)
  Role Functioning Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Role Functioning Cycle 5 Day 1 | -11.57 (21.76) | -7.22 (21.30)
  Social Functioning Cycle 2 Day 1 | -2.05 (26.92) | 0.00 (23.34)
  Social Functioning Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Social Functioning Cycle 3 Day 1 | -2.17 (23.99) | -3.49 (26.11)
  Social Functioning Cycle 4 Day 1: number analyzed (Participants) | 49 | 40
  Social Functioning Cycle 4 Day 1 | -7.14 (27.00) | -5.83 (23.74)
  Social Functioning Cycle 5 Day 1: number analyzed (Participants) | 35 | 30
  Social Functioning Cycle 5 Day 1 | -4.76 (31.72) | -9.44 (24.24)
  Insomnia Cycle 2 Day 1 | 2.92 (31.67) | -5.03 (24.80)
  Insomnia Cycle 3 Day 1: number analyzed (Participants) | 46 | 43
  Insomnia Cycle 3 Day 1 | 2.90 (25.17) | -3.10 (25.00)
  Insomnia Cycle 4 Day 1: number analyzed (Participants) | 46 | 43
  Insomnia Cycle 4 Day 1 | 7.48 (28.27) | 5.83 (31.02)
  Insomnia Cycle 5 Day 1: number analyzed (Participants) | 36 | 30
  Insomnia Cycle 5 Day 1 | 1.85 (34.68) | -5.56 (29.14)

20. Secondary Outcome: PRO Measure: Percentage of Participants With Improved, Worsened, or Remained Stable for Bothersome Side Effects of Treatment Measured by the Scales of the EORTC QLQ-C30
Description: Subjects reporting >/= 10-point increase compared to baseline (Cycle 1 Day 1) were considered "improved", those reporting <10-point difference were considered "remained stable", and those reporting >/=10-point decrease were considered "worsened". A change of at least 10 points from baseline is considered clinically meaningful (Osoba D, Rodrigues G, Myles J, et al. Interpreting the significance of changes in health-related quality of life score. J Clin Oncol 1998;16:139-44). Patient reported outcome measures were analyzed from baseline up to and including cycle 5. Scores from later timepoints were not analyzed due to attrition (in both arms, fewer than 50% of participants remained on treatment beyond cycle 5).
Time Frame: Baseline (Cycle 1 Day 1) up to Cycle 5 Day 1
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 57 | 53
Percentage of Participants
  Improved Appetite Loss: Cycle 2 | 10.5 | 18.9
  Maintained Appetite Loss: Cycle 2 | 64.9 | 66.0
  Worsened Appetite Loss: Cycle 2 | 24.6 | 15.1
  Improved Appetite Loss: Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Appetite Loss: Cycle 3 | 8.7 | 27.9
  Maintained Appetite Loss: Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Appetite Loss: Cycle 3 | 56.5 | 53.5
  Worsened Appetite Loss: Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Appetite Loss: Cycle 3 | 34.8 | 18.6
  Improved Appetite Loss: Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Appetite Loss: Cycle 4 | 10.2 | 30.0
  Maintained Appetite Loss: Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Appetite Loss: Cycle 4 | 65.3 | 57.5
  Worsened Appetite Loss: Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Appetite Loss: Cycle 4 | 24.5 | 12.5
  Improved Appetite Loss: Cycle 5: number analyzed (Participants) | 35 | 30
  Improved Appetite Loss: Cycle 5 | 8.6 | 26.7
  Maintained Appetite Loss: Cycle 5: number analyzed (Participants) | 35 | 30
  Maintained Appetite Loss: Cycle 5 | 80.0 | 53.3
  Worsened Appetite Loss: Cycle 5: number analyzed (Participants) | 35 | 30
  Worsened Appetite Loss: Cycle 5 | 11.4 | 20.0
  Improved Diarrhea: Cycle 2 | 3.5 | 7.5
  Maintained Diarrhea: Cycle 2 | 50.9 | 79.2
  Worsened Diarrhea: Cycle 2 | 45.6 | 13.2
  Improved Diarrhea: Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Diarrhea: Cycle 3 | 8.7 | 9.3
  Maintained Diarrhea: Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Diarrhea: Cycle 3 | 39.1 | 69.8
  Worsened Diarrhea: Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Diarrhea: Cycle 3 | 52.2 | 20.9
  Improved Diarrhea: Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Diarrhea: Cycle 4 | 10.2 | 10.0
  Maintained Diarrhea: Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Diarrhea: Cycle 4 | 38.8 | 77.5
  Worsened Diarrhea: Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Diarrhea: Cycle 4 | 51.0 | 12.5
  Improved Diarrhea: Cycle 5: number analyzed (Participants) | 35 | 30
  Improved Diarrhea: Cycle 5 | 14.3 | 10.0
  Maintained Diarrhea: Cycle 5: number analyzed (Participants) | 35 | 30
  Maintained Diarrhea: Cycle 5 | 34.3 | 76.7
  Worsened Diarrhea: Cycle 5: number analyzed (Participants) | 35 | 30
  Worsened Diarrhea: Cycle 5 | 51.4 | 13.3
  Improved Fatigue: Cycle 2 | 21.1 | 34.0
  Maintained Fatigue: Cycle 2 | 29.85 | 30.2
  Worsened Fatigue: Cycle 2 | 49.1 | 35.8
  Improved Fatigue: Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Fatigue: Cycle 3 | 23.9 | 34.9
  Maintained Fatigue: Cycle 3 | 15.2 | 30.2
  Worsened Fatigue: Cycle 3 | 60.9 | 34.9
  Improved Fatigue: Cycle 4: number analyzed (Participants) | 46 | 43
  Improved Fatigue: Cycle 4 | 24.5 | 28.2
  Maintained Fatigue: Cycle 4: number analyzed (Participants) | 46 | 43
  Maintained Fatigue: Cycle 4 | 28.6 | 28.2
  Worsened Fatigue: Cycle 4: number analyzed (Participants) | 46 | 43
  Worsened Fatigue: Cycle 4 | 46.9 | 43.6
  Improved Fatigue: Cycle 5: number analyzed (Participants) | 46 | 43
  Improved Fatigue: Cycle 5 | 20.0 | 30.0
  Maintained Fatigue: Cycle 5: number analyzed (Participants) | 46 | 43
  Maintained Fatigue: Cycle 5 | 20.0 | 43.3
  Worsened Fatigue: Cycle 5: number analyzed (Participants) | 46 | 43
  Worsened Fatigue: Cycle 5 | 60.0 | 26.7
  Improved Nausea/Vomiting Cycle 2 | 3.5 | 11.3
  Maintained Nausea/Vomiting Cycle 2 | 61.4 | 64.2
  Worsened Nausea/Vomiting Cycle 2 | 35.1 | 24.5
  Improved Nausea/Vomiting Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Nausea/Vomiting Cycle 3 | 4.3 | 9.3
  Maintained Nausea/Vomiting Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Nausea/Vomiting Cycle 3 | 65.2 | 62.8
  Worsened Nausea/Vomiting Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Nausea/Vomiting Cycle 3 | 30.4 | 27.9
  Improved Nausea/Vomiting Cycle 4: number analyzed (Participants) | 49 | 39
  Improved Nausea/Vomiting Cycle 4 | 2.0 | 7.5
  Maintained Nausea/Vomiting Cycle 4: number analyzed (Participants) | 49 | 39
  Maintained Nausea/Vomiting Cycle 4 | 73.5 | 67.5
  Worsened Nausea/Vomiting Cycle 4: number analyzed (Participants) | 49 | 39
  Worsened Nausea/Vomiting Cycle 4 | 24.5 | 25.0
  Improved Nausea/Vomiting Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Nausea/Vomiting Cycle 5 | 0 | 16.7
  Maintained Nausea/Vomiting Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Nausea/Vomiting Cycle 5 | 77.8 | 60.0
  Worsened Nausea/Vomiting Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Nausea/Vomiting Cycle 5 | 22.2 | 23.3
  Improved Cognitive Functioning Cycle 2 | 22.8 | 17.0
  Maintained Cognitive Function Cycle 2 | 61.4 | 60.4
  Worsened Cognitive Function Cycle 2 | 15.8 | 22.6
  Improved Cognitive Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Cognitive Functioning Cycle 3 | 26.1 | 16.3
  Maintained Cognitive Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Cognitive Functioning Cycle 3 | 47.8 | 53.5
  Worsened Cognitive Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Cognitive Functioning Cycle 3 | 26.1 | 30.2
  Improved Cognitive Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Cognitive Functioning Cycle 4 | 20.4 | 22.5
  Maintained Cognitive Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Cognitive Functioning Cycle 4 | 51.0 | 52.5
  Worsened Cognitive Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Cognitive Functioning Cycle 4 | 28.6 | 25.0
  Improved Cognitive Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Cognitive Functioning Cycle 5 | 19.4 | 20.0
  Maintained Cognitive Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Cognitive Functioning Cycle 5 | 58.3 | 46.7
  Worsened Cognitive Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Cognitive Functioning Cycle 5 | 22.2 | 33.3
  Improved Constipation Cycle 2 | 8.8 | 17.0
  Maintained Constipation Cycle 2 | 73.7 | 64.2
  Worsened Constipation Cycle 2 | 17.5 | 18.9
  Improved Constipation Cycle 3: number analyzed (Participants) | 46 | 42
  Improved Constipation Cycle 3 | 10.9 | 9.5
  Maintained Constipation Cycle 3: number analyzed (Participants) | 46 | 42
  Maintained Constipation Cycle 3 | 71.7 | 71.4
  Worsened Constipation Cycle 3: number analyzed (Participants) | 46 | 42
  Worsened Constipation Cycle 3 | 17.4 | 19.0
  Improved Constipation Cycle 4: number analyzed (Participants) | 48 | 40
  Improved Constipation Cycle 4 | 10.4 | 15.0
  Maintained Constipation Cycle 4: number analyzed (Participants) | 48 | 40
  Maintained Constipation Cycle 4 | 75.0 | 60.0
  Worsened Constipation Cycle 4: number analyzed (Participants) | 48 | 40
  Worsened Constipation Cycle 4 | 14.6 | 25.0
  Improved Constipation Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Constipation Cycle 5 | 5.6 | 13.3
  Maintained Constipation Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Constipation Cycle 5 | 80.6 | 73.3
  Worsened Constipation Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Constipation Cycle 5 | 13.9 | 13.3
  Improved Dyspnea Cycle 2: number analyzed (Participants) | 57 | 52
  Improved Dyspnea Cycle 2 | 5.3 | 15.4
  Maintained Dyspnea Cycle 2: number analyzed (Participants) | 57 | 52
  Maintained Dyspnea Cycle 2 | 77.2 | 69.2
  Worsened Dyspnea Cycle 2: number analyzed (Participants) | 57 | 52
  Worsened Dyspnea Cycle 2 | 17.5 | 15.4
  Improved Dyspnea Cycle 3: number analyzed (Participants) | 46 | 41
  Improved Dyspnea Cycle 3 | 6.5 | 14.6
  Maintained Dyspnea Cycle 3: number analyzed (Participants) | 46 | 41
  Maintained Dyspnea Cycle 3 | 67.4 | 68.3
  Worsened Dyspnea Cycle 3: number analyzed (Participants) | 46 | 41
  Worsened Dyspnea Cycle 3 | 26.1 | 17.1
  Improved Dyspnea Cycle 4: number analyzed (Participants) | 49 | 39
  Improved Dyspnea Cycle 4 | 10.2 | 12.8
  Maintained Dyspnea Cycle 4: number analyzed (Participants) | 49 | 39
  Maintained Dyspnea Cycle 4 | 69.4 | 61.5
  Worsened Dyspnea Cycle 4: number analyzed (Participants) | 49 | 39
  Worsened Dyspnea Cycle 4 | 20.4 | 25.6
  Improved Dyspnea Cycle 5: number analyzed (Participants) | 36 | 28
  Improved Dyspnea Cycle 5 | 8.3 | 14.3
  Maintained Dyspnea Cycle 5: number analyzed (Participants) | 36 | 28
  Maintained Dyspnea Cycle 5 | 69.4 | 60.7
  Worsened Dyspnea Cycle 5: number analyzed (Participants) | 36 | 28
  Worsened Dyspnea Cycle 5 | 22.2 | 25.0
  Improved Emotional Functioning Cycle 2 | 50.9 | 35.8
  Maintained Emotional Functioning Cycle 2 | 43.9 | 50.9
  Worsened Emotional Functioning Cycle 2 | 5.3 | 13.2
  Improved Emotional Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Emotional Functioning Cycle 3 | 45.7 | 37.2
  Maintained Emotional Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Emotional Functioning Cycle 3 | 45.7 | 41.9
  Worsened Emotional Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Emotional Functioning Cycle 3 | 8.7 | 20.9
  Improved Emotional Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Emotional Functioning Cycle 4 | 42.9 | 30.0
  Maintained Emotional Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Emotional Functioning Cycle 4 | 49.0 | 45.0
  Worsened Emotional Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Emotional Functioning Cycle 4 | 8.2 | 25.0
  Improved Emotional Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Improved Emotional Functioning Cycle 5 | 42.9 | 36.7
  Maintained Emotional Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Maintained Emotional Functioning Cycle 5 | 48.6 | 36.7
  Worsened Emotional Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Worsened Emotional Functioning Cycle 5 | 8.6 | 26.7
  Improved Financial Difficulties Cycle 2: number analyzed (Participants) | 56 | 52
  Improved Financial Difficulties Cycle 2 | 10.7 | 13.5
  Maintained Financial Difficulties Cycle 2: number analyzed (Participants) | 56 | 52
  Maintained Financial Difficulties Cycle 2 | 73.2 | 73.1
  Worsened Financial Difficulties Cycle 2: number analyzed (Participants) | 56 | 52
  Worsened Financial Difficulties Cycle 2 | 16.1 | 13.5
  Improved Financial Difficulties Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Financial Difficulties Cycle 3 | 13.0 | 18.6
  Maintained Financial Difficulties Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Financial Difficulties Cycle 3 | 73.9 | 72.1
  Worsened Financial Difficulties Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Financial Difficulties Cycle 3 | 13.0 | 9.3
  Improved Financial Difficulties Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Financial Difficulties Cycle 4 | 10.2 | 17.5
  Maintained Financial Difficulties Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Financial Difficulties Cycle 4 | 73.5 | 70.0
  Worsened Financial Difficulties Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Financial Difficulties Cycle 4 | 16.3 | 12.5
  Improved Financial Difficulties Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Financial Difficulties Cycle 5 | 13.9 | 20.0
  Maintained Financial Difficulties Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Financial Difficulties Cycle 5 | 66.7 | 63.3
  Worsened Financial Difficulties Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Financial Difficulties Cycle 5 | 19.4 | 16.7
  Improved Pain Cycle 2 | 35.1 | 35.8
  Maintained Pain Cycle 2 | 40.4 | 45.3
  Worsened Pain Cycle 2 | 24.6 | 18.9
  Improved Pain Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Pain Cycle 3 | 37.0 | 39.5
  Maintained Pain Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Pain Cycle 3 | 39.1 | 39.5
  Worsened Pain Cycle: number analyzed (Participants) | 46 | 43
  Worsened Pain Cycle | 23.9 | 20.9
  Improved Pain Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Pain Cycle 4 | 32.7 | 37.5
  Maintained Pain Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Pain Cycle 4 | 32.7 | 35.0
  Worsened Pain Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Pain Cycle 4 | 34.7 | 27.5
  Improved Pain Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Pain Cycle 5 | 33.3 | 33.3
  Maintained Pain Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Pain Cycle 5 | 30.6 | 40.0
  Worsened Pain Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Pain Cycle 5 | 36.1 | 26.7
  Improved Physical Functioning Cycle 2 | 7.0 | 13.2
  Maintained Physical Functioning Cycle 2 | 68.4 | 75.5
  Worsened Physical Functioning Cycle 2 | 24.6 | 11.3
  Improved Physical Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Physical Functioning Cycle 3 | 8.7 | 16.3
  Maintained Physical Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Physical Functioning Cycle 3 | 67.4 | 60.5
  Worsened Physical Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Physical Functioning Cycle 3 | 23.9 | 23.3
  Improved Physical Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Physical Functioning Cycle 4 | 4.1 | 17.5
  Maintained Physical Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Physical Functioning Cycle 4 | 55.1 | 57.5
  Worsened Physical Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Physical Functioning Cycle 4 | 40.8 | 25.0
  Improved Physical Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Physical Functioning Cycle 5 | 8.3 | 16.7
  Maintained Physical Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Physical Functioning Cycle 5 | 44.4 | 46.7
  Worsened Physical Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Physical Functioning Cycle 5 | 47.2 | 36.7
  Improved Global Health Status/QoL Cycle 2 | 19.3 | 26.4
  Maintained Global Health Status/QoL Cycle 2 | 45.6 | 58.5
  Worsened Global Health Status/QoL Cycle 2 | 35.1 | 15.1
  Improved Global Health Status/QoL Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Global Health Status/QoL Cycle 3 | 17.4 | 25.6
  Maintained Global Health Status/QoL Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Global Health Status/QoL Cycle 3 | 37.0 | 60.5
  Worsened Global Health Status/QoL Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Global Health Status/QoL Cycle 3 | 45.7 | 14.0
  Improved Global Health Status/QoL Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Global Health Status/QoL Cycle 4 | 14.3 | 25.0
  Maintained Global Health Status/QoL Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Global Health Status/QoL Cycle 4 | 51.0 | 42.5
  Worsened Global Health Status/QoL Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Global Health Status/QoL Cycle 4 | 34.7 | 32.5
  Improved Global Health Status/QoL Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Global Health Status/QoL Cycle 5 | 11.1 | 20.0
  Maintained Global Health Status/QoL Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Global Health Status/QoL Cycle 5 | 58.3 | 46.7
  Worsened Global Health Status/QoL Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Global Health Status/QoL Cycle 5 | 30.6 | 33.3
  Improved Role Functioning Cycle 2 | 17.5 | 24.5
  Maintained Role Functioning Cycle 2 | 52.6 | 45.3
  Worsened Role Functioning Cycle 2 | 29.8 | 30.2
  Improved Role Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Role Functioning Cycle 3 | 13.0 | 27.9
  Maintained Role Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Role Functioning Cycle 3 | 47.8 | 46.5
  Worsened Role Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Role Functioning Cycle 3 | 39.1 | 25.6
  Improved Role Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Role Functioning Cycle 4 | 12.2 | 25.0
  Maintained Role Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Role Functioning Cycle 4 | 38.8 | 37.5
  Worsened Role Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Role Functioning Cycle 4 | 49.0 | 37.5
  Improved Role Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Improved Role Functioning Cycle 5 | 11.1 | 16.7
  Maintained Role Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Maintained Role Functioning Cycle 5 | 47.2 | 40.0
  Worsened Role Functioning Cycle 5: number analyzed (Participants) | 36 | 30
  Worsened Role Functioning Cycle 5 | 41.7 | 43.3
  Improved Social Functioning Cycle 2 | 21.1 | 22.6
  Maintained Social Functioning Cycle 2 | 49.1 | 49.1
  Worsened Social Functioning Cycle 2 | 29.8 | 28.3
  Improved Social Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Improved Social Functioning Cycle 3 | 17.4 | 16.3
  Maintained Social Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Maintained Social Functioning Cycle 3 | 52.2 | 53.5
  Worsened Social Functioning Cycle 3: number analyzed (Participants) | 46 | 43
  Worsened Social Functioning Cycle 3 | 30.4 | 30.2
  Improved Social Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Improved Social Functioning Cycle 4 | 16.3 | 10.0
  Maintained Social Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Maintained Social Functioning Cycle 4 | 49.0 | 47.5
  Worsened Social Functioning Cycle 4: number analyzed (Participants) | 49 | 40
  Worsened Social Functioning Cycle 4 | 34.7 | 42.5
  Improved Social Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Improved Social Functioning Cycle 5 | 17.1 | 13.3
  Maintained Social Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Maintained Social Functioning Cycle 5 | 48.6 | 36.7
  Worsened Social Functioning Cycle 5: number analyzed (Participants) | 35 | 30
  Worsened Social Functioning Cycle 5 | 34.3 | 50.0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug or until initiation of another anti-cancer therapy, whichever occurs first (up to 3 years, 3 months)
Arm/Group | Ipatasertib and Paclitaxel | Placebo and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 41/61 | 46/62
Serious Adverse Events (participants affected / at risk) | 18/61 | 12/62
Other Adverse Events (participants affected / at risk) | 61/61 | 59/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipatasertib and Paclitaxel (N=61) | Placebo and Paclitaxel (N=62)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Retroperitoneal Infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0)
Cell Death (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipatasertib and Paclitaxel (N=61) | Placebo and Paclitaxel (N=62)
Anxiety (Psychiatric disorders) | 2 (3) | 4 (6)
Insomnia (Psychiatric disorders) | 13 (19) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 8 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 33 (37) | 29 (34)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 10 (17) | 5 (5)
Nail Disorder (Skin and subcutaneous tissue disorders) | 4 (7) | 4 (4)
Onycholysis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (14) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 17 (28) | 13 (17)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7)
Flushing (Vascular disorders) | 4 (4) | 3 (3)
Hot Flush (Vascular disorders) | 5 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (12) | 5 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (15) | 4 (10)
Urinary Tract Infection (Infections and infestations) | 5 (6) | 4 (4)
Alanine Aminotransferase Increased (Investigations) | 3 (5) | 4 (4)
Aspartate Aminotransferase Increased (Investigations) | 5 (8) | 3 (6)
Neutrophil Count Decreased (Investigations) | 8 (19) | 9 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 6 (7)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (9) | 4 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (42) | 15 (25)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 2 (2)
Dizziness (Nervous system disorders) | 11 (19) | 9 (10)
Dysgeusia (Nervous system disorders) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 11 (15) | 13 (14)
Hypoaesthesia (Nervous system disorders) | 4 (6) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 12 (17) | 14 (18)
Paraesthesia (Nervous system disorders) | 6 (10) | 7 (10)
Peripheral Sensory Neuropathy (Nervous system disorders) | 16 (33) | 10 (16)
Anaemia (Blood and lymphatic system disorders) | 9 (17) | 8 (11)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 13 (38) | 15 (36)
Abdominal Pain (Gastrointestinal disorders) | 9 (13) | 7 (9)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 4 (5)
Constipation (Gastrointestinal disorders) | 12 (17) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 56 (205) | 13 (19)
Dry Mouth (Gastrointestinal disorders) | 2 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (11) | 6 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastritis (Gastrointestinal disorders) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 32 (67) | 21 (28)
Stomatitis (Gastrointestinal disorders) | 11 (14) | 5 (6)
Vomiting (Gastrointestinal disorders) | 17 (39) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 5 (6)
Asthenia (General disorders) | 17 (41) | 7 (7)
Chest Discomfort (General disorders) | 4 (4) | 1 (1)
Chest Pain (General disorders) | 4 (5) | 6 (6)
Fatigue (General disorders) | 18 (26) | 20 (32)
Mucosal Inflammation (General disorders) | 4 (7) | 4 (5)
Oedema Peripheral (General disorders) | 7 (9) | 5 (6)
Pyrexia (General disorders) | 11 (13) | 7 (9)
Dry Eye (Eye disorders) | 4 (5) | 3 (3)
Influenza (Infections and infestations) | 4 (6) | 1 (1)
Rhinitis (Infections and infestations) | 4 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 12 (15) | 11 (15)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (10) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.